CLINICAL TRIAL: NCT02375880
Title: A Dose Escalation and Cohort Expansion Study of DKN-01 in Combination With Gemcitabine and Cisplatin in Patients With Advanced Carcinoma Primary to the Intra- or Extra-hepatic Biliary System or Gallbladder
Brief Title: Study of DKN-01 and Gemcitabine/Cisplatin in Patients With Carcinoma to Primary to the Intra- or Extra-Hepatic Biliary System or Gallbladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEK-DKK1-P103
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma of Intrahepatic and Extra-hepatic Biliary System; Carcinoma of Gallbladder; Bile Duct Cancer; Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Bile Duct Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 150 mg DKN-01 Part A (Experimental): Patients will receive 150 mg of DKN-01 followed by gemcitabine 1000 mg/m2 and cisplatin 25 mg/m2 on Days 1 and 8 of each 21-day cycle.
  Interventions: Drug: DKN-01; Drug: gemcitabine; Drug: cisplatin
- 300 mg DKN-01 Part A (Experimental): Patients will receive 300 mg of DKN-01 followed by gemcitabine 1000 mg/m2 and cisplatin 25 mg/m2 on Days 1 and 8 of each 21-day cycle.
  Interventions: Drug: DKN-01; Drug: gemcitabine; Drug: cisplatin
- MTD mg DKN-01 Part B (Experimental): Patients are treated at the maximum tolerated dose (MTD) of DKN-01 (or highest dose tested in Part A if the MTD is not defined) followed by gemcitabine 1000 mg/m2 and cisplatin 25 mg/m2 on Days 1 and 8 of each 21-day cycle.
  Interventions: Drug: DKN-01; Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: DKN-01 — Administration by intravenous (IV) infusion.
  Other Names: LY2812176
Drug: gemcitabine — Administered by IV infusion.
  Other Names: Gemzar
Drug: cisplatin — Administered by IV infusion
  Other Names: Platinol

SUMMARY:
DKN-01 is a humanized monoclonal antibody (Mab) with neutralizing activity against Dkk-1 and is being developed as an anti-neoplastic agent. This study is designed to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of DKN-01 in combination with gemcitabine and cisplatin in patients with carcinoma primary to the intra- or exta-hepatic biliary system or gallbladder.

DETAILED DESCRIPTION:
In Part A, escalating doses of DKN-01 will be administered to different cohorts of patients to evaluate safety and dose limiting toxicities (DLTs) and to establish the maximum tolerated dose of DKN-01 when administered in combination with gemcitabine and cisplatin.

Part B is an expansion cohort in which patients are treated at the MTD of DKN-01 (or highest dose tested if the MTD is not defined) to further characterize safety, tolerability, pharmacokinetics and efficacy within the defined patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has carcinoma primary to the intra- or extra-hepatic biliary system or gall bladder.
2. Patient must have sufficient tumor tissue available for submission.
3. For patients who have received prior cryotherapy, radiofrequency ablation, radioembolization, ethanol injection, transarterial chemoembolization (TACE) or photodynamic therapy, at least 28 days must have elapsed since that therapy, and lesions that have not been treated with local therapy must be present and measurable.
4. Patients may have received prior adjuvant chemotherapy with gemcitabine with or without cisplatin, as long as 6 months have elapsed since last treatment.
5. Patients must have one or more tumors measurable on radiographic imaging as defined by RECIST.
6. ECOG PS of 0 or 1. Patients with an ECOG PS of 2 may be entered upon review and approval of the medical monitor.
7. Estimated life expectancy of at least 3 months.
8. Disease-free of active second/secondary or prior malignancies for ≥ 2 years with the exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or breast.
9. Adequate hematological, renal, hepatic and coagulation laboratory test results.
10. Women of child bearing potential and men must agree to use adequate contraception during the study and for 6 months after their last dose of study drug.
11. Available for the duration of the study and are willing to follow study-specific procedures.
12. Provide written informed consent

Exclusion Criteria:

1. New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, or unstable arrhythmia.
2. Have Fridericia-corrected QT interval (QTcF) > 470 msec (female) or > 450 (male), or history of congenital long QT syndrome.
3. Active, uncontrolled bacterial, viral, or fungal infections.
4. Known to be human immunodeficiency virus (HIV) positive or has untreated, active hepatitis B.
5. History of major organ transplant.
6. History of an autologous/allogenic bone marrow transplant.
7. Serious nonmalignant disease.
8. Pregnant or nursing.
9. History of osteonecrosis of the hip or have evidence of structural bone abnormalities in the proximal femur on MRI scan that are symptomatic and clinically significant.
10. Symptomatic central nervous system (CNS) malignancy or metastasis.
11. Clinically significant peripheral neuropathy
12. Known osteoblastic bony metastasis.
13. Treatment with surgery or chemotherapy within 21 days prior to study entry or radiation within 14 days of study entry.
14. Previously treated with an anti-Dkk-1 therapy.
15. Other exclusions apply

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-06; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose-limiting toxicities as determined in Part A. | End of Cycle 1 (Day 21)
  Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v 4.03).
Composite Safety parameters as assessed by new or changing physical examinations, vital signs, electrocardiograms (ECGs), clinical laboratories, concomitant medication reviews, and assessment of adverse events. | Parts A and B: at a minimum Days 1, 8, 15 of each treatment cycle.

SECONDARY OUTCOMES:
Pharmacokinetics - AUC | Cycle 1 - Days 1 and 8, Cycle 2 - Day 1
  Plasma levels will be measured during the treatment period.
Pharmacokinetics - Cmax | Cycle 1 - Days 1 and 8, Cycle 2 - Day 1
  Plasma levels will be measured during the treatment period.
Pharmacokinetics - Tmax | Cycle 1 - Days 1 and 8, Cycle 2 - Day 1
  Plasma levels will be measured during the treatment period.
Efficacy - Response to treatment evaluated using the Response Evaluation Criteria in Solid Tumors guidelines (RECIST 1.1) | At baseline, prior to the start of Cycle 3, and every 2 cycles thereafter until disease progression or death
  Response to treatment evaluated using the Response Evaluation Criteria in Solid Tumors guidelines (RECIST 1.1).

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - University Hospitals, Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Goyal L, Sirard C, Schrag M, Kagey MH, Eads JR, Stein S, El-Khoueiry AB, Manji GA, Abrams TA, Khorana AA, Miksad R, Mahalingam D, Zhu AX, Duda DG. Phase I and Biomarker Study of the Wnt Pathway Modulator DKN-01 in Combination with Gemcitabine/Cisplatin in Advanced Biliary Tract Cancer. Clin Cancer Res. 2020 Dec 1;26(23):6158-6167. doi: 10.1158/1078-0432.CCR-20-1310. Epub 2020 Sep 2. PMID 32878766